CLINICAL TRIAL: NCT04499261
Title: A Prospective Cohort Study: Laparoscopic Versus Open Surgery for Lesions Originating in the Paracaval Portion of the Caudate Lobe
Brief Title: Laparoscopic Versus Open Surgery for Lesions Originating in the Paracaval Portion of the Caudate Lobe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHZSG010
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Paracaval Portion
Keywords: Laparoscopy; hepatectomy; Caudate Lobe
MeSH Terms: interventions — Laparoscopy; Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic surgery (Experimental): The laparoscopic view is caudal to cephalic, which is consistent with the direction of hepatic transection. In addition, the high-definition magnified view and ability to change perspectives with the laparoscope are conducive to subtle manipulation, and compression of the carbon dioxide pneumoperitoneum can reduce venous bleeding. Therefore, laparoscopic surgery may have certain advantages in the treatment of paracaval-originating lesions.
  Interventions: Procedure: laparoscopic surgery
- Open surgery (Active Comparator): Open surgery is the traditional surgical method for resection of paracaval-originating lesions.
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — Patients were supine in a reverse Trendelenburg position and received intravenous inhalation combined with anesthesia. The patients' legs were spread apart. A carbon dioxide pneumoperitoneum was established. The intermittent Pringle's maneuver was carried out when necessary. Five trocars were placed in a fan shape around the lesion. Cholecystectomy was performed routinely. First, the liver was mobilized. Then, the liver parenchyma was transected and the branches of the hepatic veins and pedicles encountered were clipped and divided. The lesion was meticulously separated from the vascular structures and liver parenchyma and completely resected. The raw surface was treated with bipolar coagulation to achieve hemostasis and repeatedly washed until no bleeding or bile leakage was confirmed. Finally, the specimens were packed in a specimen bag and removed. The raw surface was packed with biological hemostatic materials, and drainage tubes were routinely placed.
  Arms: laparoscopic surgery
Procedure: Open surgery — Patients were placed in the supine position and received intravenous inhalation combined with anesthesia. The intermittent Pringle's maneuver was carried out when necessary. Routinely, a reversed L-shape incision was performed. Cholecystectomy was performed routinely. First, the liver was mobilized. Then, the liver parenchyma was transected and the branches of the hepatic veins and pedicles encountered were clipped and divided. The lesion was meticulously separated from the vascular structures and liver parenchyma and completely resected. The raw surface was treated with bipolar coagulation to achieve hemostasis and repeatedly washed until no bleeding or bile leakage was confirmed. Finally, the specimens were packed in a specimen bag and removed. The raw surface was packed with biological hemostatic materials, and drainage tubes were routinely placed.
  Arms: Open surgery

SUMMARY:
This study aimed to evaluate the safety, feasibility and efficacy of laparoscopic for resecting paracaval-originating lesions by contrast of open procedures.

DETAILED DESCRIPTION:
The paracaval portion of the caudate lobe is located in the core of the liver. Lesions originating in the paracaval portion often cling to or even invade major hepatic vascular structures. Open surgery is the traditional surgical method for resection of paracaval-originating lesions. With the development of laparoscopic surgery, paracaval-originating lesions are no longer an absolute contraindication for laparoscopic procedures. The high-definition magnified view and ability to change perspectives with the laparoscope are conducive to subtle manipulation, and compression of the carbon dioxide pneumoperitoneum can reduce venous bleeding. Nevertheless, laparoscopic anterior hepatic transection for paracaval-originating lesion resection is still a challenging procedure, and only a few cases have been reported. This study aimed to evaluate the safety, feasibility and efficacy of laparoscopic for resecting paracaval-originating lesions by contrast of open procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Between 18 to 70 years, both male and female
2. The general condition of the patient can tolerate anesthesia and surgery
3. Paracaval-originating lesion diagnosis is clear preoperative
4. No rupture of the tumor, no bloody ascites, no invasion of the surrounding tissues and distant metastasis
5. Liver function ≥ Child-pugh level B, indocyanine green retention rate at 15 min ≤ 15%, the residual liver volume and standard liver volume ratio ≥ 40%.
6. Upper abdominal surgery, radiofrequency ablation, Transhepatic Arterial Chemotherapy And Embolization treatment, radiotherapy and chemotherapy have not been implemented
7. Volunteer to participate in the study and sign informed consent

Exclusion Criteria:

1. Age:Younger than 18 or more than 70 years old 2. Pregnant and lactating women 3. Severe cirrhosis, portal hypertension, or active hepatitis are present 4. Severe upper abdominal adhesions 5. The lesion originated in other parts of the liver other than the paracaval portion 6. Patients with poor general condition and could not tolerate surgery or anesthesia

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-09-25 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
survival rate | 3 years
  follow-up after the surgery every 3months, to understand relapse, death, statistics 1-year, 3-year overall survival rates，disease-free survival rates , recurrence and metastasis rate.

SECONDARY OUTCOMES:
operation time | during the operation
  intraoperative parameter
intraoperative blood loss | during the operation
  intraoperative parameter
rate of blood transfusion. | during the operation
  intraoperative parameter

OTHER OUTCOMES:
postoperative complications | Duration hospitalization(an expected average of 7 days)
  ascites, pleural effusion,cardiopulmonary insufficiency,mortality, postoperative liver function failure.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, M.D., Study Director — Shuguo Zheng, MD Study Director Institute of Hepatobiliary Surgery, Southwest Hospital, Army medical university
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China